CLINICAL TRIAL: NCT05207735
Title: Henan Cancer Hospital, Affiliated Cancer Hospital of Zhengzhou University.
Brief Title: PD-1 Inhibitor Sintilimab Combined With Capecitabine for Adjuvant Treatment After Radical Resection of Cholangiocarcinoma.
Acronym: SCRCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-246
Record Dates: First submitted 2021-11-24; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Cholangiocarcinoma
Keywords: PD-1 Inhibitor; Capecitabine; Adjuvant Treatment
MeSH Terms: conditions — Cholangiocarcinoma | interventions — sintilimab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GROUP 1 (Experimental): Sintilizumab, 200 mg, intravenous infusion, a treatment cycle every 3 weeks, administration on the first day of each cycle, 6 cycles.
  Capecitabine: 1250 mg/m2, orally, twice a day, 1-14 days, one treatment cycle every three weeks, 8 cycles.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — * Sintilizumab, 200 mg, intravenous infusion, a treatment cycle every 3 weeks, administration on the first day of each cycle, 6 cycles.
  * Capecitabine: 1250 mg/m2, orally, twice a day, 1-14 days, one treatment cycle every three weeks, 8 cycles.
  Other Names: Capecitabine

SUMMARY:
This is a single-center, single-arm, prospective phase II clinical study to evaluate the effectiveness and safety of Sintilimab combined with capecitabine in patients after radical resection of cholangiocarcinoma.

The primary endpoint of the study:

• 2-year recurrence-free survival rate

Secondary endpoint:

• Overall survival (OS), 1y RFS%, 2y OS%, 3y OS%, time to recurrence (TTR), RFS;Safety and tolerability.

Study drugs, dosages, and methods of administration:

* Sintilizumab, 200 mg, intravenous infusion, a treatment cycle every 3 weeks, administration on the first day of each cycle, 6 cycles.
* Capecitabine: 1250 mg/m2, orally, twice a day, 1-14 days, one treatment cycle every three weeks, 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18-75 years old;
2. Sign written informed consent, and be able to comply with the visits and related procedures stipulated in the plan;
3. Histopathological diagnosis was extrahepatic cholangiocarcinoma, including hilar cholangiocarcinoma and distal cholangiocarcinoma, and had undergone radical resection;
4. The pathology report of the patient must confirm complete resection (recovery from the operation to be disease-free, and the sample has negative margins R0, R1);
5. The patient must be treated within 12 weeks after the radical resection;
6. No anti-tumor treatment before radical resection, including radiotherapy and chemotherapy, targeted therapy and immunotherapy;
7. ECOG score 0-1 points;
8. Expected survival time> 6 months;
9. With sufficient organ and bone marrow function, the laboratory test values within 7 days before randomization meet the following requirements (no blood components, cell growth factors, albumin and other corrective treatment drugs are allowed to meet the conditions), as follows :1) Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L; platelet count (platelet, PLT) ≥75×10 9/L; hemoglobin content (hemoglobin, HGB) ≥9.0 g /dL;2) Liver function: serum total bilirubin (TBIL) ≤ 2×upper limit of normal value (ULN); alanine aminotransferase (ALT) and aspartate amino transfer Enzyme (aspartate transferase, AST) ≤5×ULN; serum albumin ≥28 g/L; alkaline phosphatase (alkaline phosphatase, ALP) ≤5×ULN;3) Renal function: serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance (clearance of creatinine, CCr) ≥ 50 mL/min (Cockcroft-Gault formula); urine routine results show urine protein <2+; against baseline For patients whose urine protein is ≥2+ by routine urine test, 24-hour urine collection and 24-hour urine protein quantitative <1g should be performed;4) Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
10. Female patients of childbearing age or male patients whose sexual partners are females of childbearing age should take effective contraceptive measures throughout the treatment period and 6 months after the last treatment.

Exclusion Criteria:

1. Diagnosis of other malignant diseases outside the biliary tract within 5 years before the first administration (excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma, and/or radically excised carcinoma in situ);
2. Currently participating in interventional clinical research treatment, or received other research drugs or used research devices within 4 weeks before the first administration;
3. Have received the following therapies in the past: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or for another stimulating or synergistic inhibition of T cell receptors (for example, CTLA-4, OX-40, CD137) drug;
4. Have received radiotherapy for biliary tract tumors in the past;
5. Received Chinese patent medicines with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural effusion) systemic systemic treatment within 2 weeks before the first administration;
6. An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatments. Known history of primary immunodeficiency. Only patients with positive autoimmune antibodies need to confirm whether there are autoimmune diseases based on the judgment of the investigator;
7. Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy within 4 weeks before the first administration of the study. Note: Physiological doses of glucocorticoids are allowed (≤10 mg/day prednisone or equivalent drugs);
8. There is clinically uncontrollable pleural effusion/abdominal effusion (patients who do not need to drain the effusion or stop drainage for 3 days without a significant increase in effusion can be included in the group)
9. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
10. Those who are known to be allergic to the active ingredients or excipients of Sintilimab
11. Before starting treatment, have not fully recovered from toxicity and/or complications caused by any intervention (ie, ≤ Grade 1 or reached baseline, excluding fatigue or hair loss)
12. Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive)
13. Untreated active hepatitis B (defined as HBsAg positive and the number of copies of HBV-DNA detected at the same time is greater than the upper limit of normal value of the laboratory department of the research center).Note: Hepatitis B subjects who meet the following criteria can also be included in the group:1) The HBV viral load before the first administration is less than 2.5×103 copies/ml (500 IU/ml), and the subject should receive anti-HBV treatment during the entire study treatment period;2) For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), there is no need to receive preventive anti-HBV treatment, but close monitoring of virus reactivation is required.
14. Active HCV infected subjects (HCV antibody-positive and HCV-RNA level is higher than the lower limit of detection);
15. Have received a live attenuated vaccine within 4 weeks before the first dose;
16. Pregnant or lactating women;
17. There are any serious or uncontrollable systemic diseases, such as:1) The resting electrocardiogram has major abnormalities in rhythm, conduction, or morphology that are severe and difficult to control, such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation;2) Unstable angina pectoris, congestive heart failure, chronic heart failure of New York Heart Association (NYHA) grade ≥ 2;3) Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, occurred within 6 months before being selected for treatment;4) Major surgery (craniotomy, thoracotomy or laparotomy) or unhealed wounds, ulcers or fractures have been received within 4 weeks before the first administration. Have received tissue biopsy or other minor surgical procedures within 7 days before the first administration, except for venipuncture catheters for the purpose of intravenous infusion;5) Unsatisfactory blood pressure control (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);6) Active tuberculosis;7) There is an active or uncontrolled infection that requires systemic treatment;8) There is clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;9) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;10) Poor control of diabetes (fasting blood glucose (FBG)> 10mmol/L);11) Urine routine test shows urine protein ≥++, and the 24-hour urine protein quantitative is confirmed to be >1.0 g;12) Patients with mental disorders who cannot cooperate with treatment;
18. The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subject from participating in the study, or the investigator believes that it is not suitable for inclusion in the group. The investigator believes that there are other potential risks and is not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
2y RFS% | up to 24 months
  2-year recurrence-free survival rate

SECONDARY OUTCOMES:
OS | up to 36 months
  overall survival
1y RFS% | up to 12 months
  1-year recurrence-free survival rate
2y OS% | up to 24 months
  2-year overall survival rate
3y OS% | up to 36 months
  3-year overall survival rate
TTR | up to 36 months
  time to recurrence
RFS | 1-36 months
  recurrence-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jinxue Zhou, MD, Study Chair — Henan cancer hospital,affiliated cancer hospital of zhengzhou university

IPD SHARING:
Plan to Share IPD: No